CLINICAL TRIAL: NCT03434249
Title: Studio Clinico Randomizzato Per Valutare l'Efficacia Del Bifidobacterium BB-12® Nel Trattamento Delle Coliche Infantili
Brief Title: Clinical Trial to Evaluate the Efficacy of Bifidobacterium BB-12® in the Treatment of Infantile Colic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SOFAR S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-DS BIGI
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Results first posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Infantile Colic; Colic, Infantile
Keywords: Bifidobacterium
MeSH Terms: conditions — Colic

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized double blind placebo controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): patients who take Bifidobacterium BB-12® (Bifidolactis Infant), 6 drops a day (guaranteeing a billion of living cells) for 28 consecutive days;
  Interventions: Dietary Supplement: Bifidobacterium, BB-12® (Bifidolactis Infant)
- Group II (Placebo Comparator): patients who take Bifidolactis Infant Placebo 6 drops a day for 28 consecutive days.
  Interventions: Dietary Supplement: Bifidolactis Infant Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium, BB-12® (Bifidolactis Infant)
  Arms: Group I
Dietary Supplement: Bifidolactis Infant Placebo
  Arms: Group II

SUMMARY:
This is a single-center, randomized, double blind controlled study to investigate the effects of Bifidobacterium, BB-12® versus placebo in a study group of pediatric patients with infantile colic.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if they meet all the following criteria:

* Exclusively breastfed healthy infants of both sexes, aged ≤ 7 weeks.
* Diagnosis of IC according to Rome III criteria.
* Written informed consent of the parent/tutor.

Exclusion Criteria:

Patients are excluded from this study if they meet any of the following criteria:

* Birth weight < 2500 g.
* Gestational age < 37 weeks.
* APGAR 5 minutes < 7.
* Formula feeding.
* Stunting/loss of weight (< 100 g/weeks from birth to the last reported weight).
* Neurological diseases.
* Known or suspected food allergy.
* Gastroesophageal reflux disease.
* Use of substances that alter gut microbiota (probiotics, prebiotics, antibiotics, gastric acidity inhibitors) in the last 2 weeks prior the enrollment.
* History of fever and/or infectious diseases in the last 2 weeks prior to enrollment.
* Ongoing systemic infections.
* History of congenital infections.
* Chronic intestinal diseases (cystic fibrosis or other forms of primitive pancreatic insufficiency)
* Primitive or secondary malformations of the gastrointestinal tract (such as esophageal atresia, intestinal atresia, short bowel syndrome, malrotation).
* Metabolic diseases.
* Genetic diseases and chromosomal abnormalities.
* Primary or secondary immunodeficiencies.
* Not sufficient reliability or presence of conditions that may result in non-compliance/adherence of the patient to the Protocol.
* Previous participation in this study.

Max Age: 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2016-11-11 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Berni Canani, Prof., Principal Investigator — Federico II University
Locations (1):
- Dipartimento di Scienze Mediche Traslazionali - Sezione Pediatria - Università degli Studi di napoli "Federico II", Napoli, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hyman PE, Milla PJ, Benninga MA, Davidson GP, Fleisher DF, Taminiau J. Childhood functional gastrointestinal disorders: neonate/toddler. Gastroenterology. 2006 Apr;130(5):1519-26. doi: 10.1053/j.gastro.2005.11.065. PMID 16678565
- [Background] Szajewska H, Gyrczuk E, Horvath A. Lactobacillus reuteri DSM 17938 for the management of infantile colic in breastfed infants: a randomized, double-blind, placebo-controlled trial. J Pediatr. 2013 Feb;162(2):257-62. doi: 10.1016/j.jpeds.2012.08.004. Epub 2012 Sep 14. PMID 22981952
- [Background] Kabeerdoss J, Devi RS, Mary RR, Prabhavathi D, Vidya R, Mechenro J, Mahendri NV, Pugazhendhi S, Ramakrishna BS. Effect of yoghurt containing Bifidobacterium lactis Bb12(R) on faecal excretion of secretory immunoglobulin A and human beta-defensin 2 in healthy adult volunteers. Nutr J. 2011 Dec 23;10:138. doi: 10.1186/1475-2891-10-138. PMID 22196482
- [Background] Mohan R, Koebnick C, Schildt J, Mueller M, Radke M, Blaut M. Effects of Bifidobacterium lactis Bb12 supplementation on body weight, fecal pH, acetate, lactate, calprotectin, and IgA in preterm infants. Pediatr Res. 2008 Oct;64(4):418-22. doi: 10.1203/PDR.0b013e318181b7fa. PMID 18552710
- [Background] Mohan R, Koebnick C, Schildt J, Schmidt S, Mueller M, Possner M, Radke M, Blaut M. Effects of Bifidobacterium lactis Bb12 supplementation on intestinal microbiota of preterm infants: a double-blind, placebo-controlled, randomized study. J Clin Microbiol. 2006 Nov;44(11):4025-31. doi: 10.1128/JCM.00767-06. Epub 2006 Sep 13. PMID 16971641
- [Background] Savino F, Cordisco L, Tarasco V, Calabrese R, Palumeri E, Matteuzzi D. Molecular identification of coliform bacteria from colicky breastfed infants. Acta Paediatr. 2009 Oct;98(10):1582-8. doi: 10.1111/j.1651-2227.2009.01419.x. Epub 2009 Jul 9. PMID 19604166
- [Background] Hall B, Chesters J, Robinson A. Infantile colic: a systematic review of medical and conventional therapies. J Paediatr Child Health. 2012 Feb;48(2):128-37. doi: 10.1111/j.1440-1754.2011.02061.x. Epub 2011 Apr 7. PMID 21470331
- [Background] Savino F, Bailo E, Oggero R, Tullio V, Roana J, Carlone N, Cuffini AM, Silvestro L. Bacterial counts of intestinal Lactobacillus species in infants with colic. Pediatr Allergy Immunol. 2005 Feb;16(1):72-5. doi: 10.1111/j.1399-3038.2005.00207.x. PMID 15693915
- [Background] Savino F, Cresi F, Pautasso S, Palumeri E, Tullio V, Roana J, Silvestro L, Oggero R. Intestinal microflora in breastfed colicky and non-colicky infants. Acta Paediatr. 2004 Jun;93(6):825-9. PMID 15244234
- [Background] Gupta SK. Is colic a gastrointestinal disorder? Curr Opin Pediatr. 2002 Oct;14(5):588-92. doi: 10.1097/00008480-200210000-00005. PMID 12352253
- [Background] Lucassen PL, Assendelft WJ, van Eijk JT, Gubbels JW, Douwes AC, van Geldrop WJ. Systematic review of the occurrence of infantile colic in the community. Arch Dis Child. 2001 May;84(5):398-403. doi: 10.1136/adc.84.5.398. PMID 11316682
- [Background] BRAZELTON TB. Crying in infancy. Pediatrics. 1962 Apr;29:579-88. No abstract available. PMID 13872677
- [Background] Iacovou M, Ralston RA, Muir J, Walker KZ, Truby H. Dietary management of infantile colic: a systematic review. Matern Child Health J. 2012 Aug;16(6):1319-31. doi: 10.1007/s10995-011-0842-5. PMID 21710185

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was a randomized, double-blind, placebo-controlled parallel-group study. Eighty (80) infants were screened and all were enrolled in the study and randomized (40 to Bifidobacteriium BB-12® and 40 to Placebo).
  The enrollment period started on 11-Nov-2016 and closed on 6-Nov-2017.
Groups:
- Bifidobacterium BB-12®: patients who take Bifidobacterium BB-12® (Bifidolactis Infant), 6 drops a day (guaranteeing a billion of living cells) for 28 consecutive days.
- Placebo: patients who take Bifidolactis Infant Placebo 6 drops a day for 28 consecutive days.
Period: Overall Study
Arm/Group | Bifidobacterium BB-12® | Placebo
Started | 40 | 40
Completed | 35 | 37
Not Completed | 5 | 3
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance of family | 2 | 1
Not completed — Difficulties in completing daily diary | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Bifidobacterium BB-12®: patients who take Bifidobacterium BB-12® (Bifidolactis Infant), 6 drops a day (guaranteeing a billion of living cells) for 28 consecutive days;
  Bifidobacterium, BB-12® (Bifidolactis Infant)
- Placebo: patients who take Bifidolactis Infant Placebo 6 drops a day for 28 consecutive days.
  Bifidolactis Infant Placebo
- Total: Total of all reporting groups
Arm/Group | Bifidobacterium BB-12® | Placebo | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: days] | 33.05 (5.03) | 32.73 (5.69) | 32.89 (5.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 22 | 21 | 43
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 40 | 40 | 80
Type of childbirth [Count of Participants; unit: Participants]
  Caesarean section | 25 | 19 | 44
  Natural childbirth | 15 | 21 | 36
Gestational age [Mean (Standard Deviation); unit: weeks] | 38.43 (0.93) | 38.53 (1.20) | 38.48 (1.07)
Birth weight [Mean (Standard Deviation); unit: grams] | 3280.75 (367.54) | 3412.00 (442.75) | 3346.38 (409.66)
Apgar 5 minutes score [Mean (Standard Deviation); unit: scores on a scale] — The Apgar score (APGAR is the acronym of Appearance, Pulse, Grimace, Activity, Respiration) is a method used to summarize the health of newborn children. It evaluates five parameters (Skin colors, Pulse rate, Reflex irritability grimace, Muscle tone, Respiratory effort) assigning to each parameter a score from 0 to 2 (values 0, 1, 2) and summing up the five values. The resulting score ranges from 0 to 10. APGAR 5 minutes means that the test is done at 5 minutes after birth. Scores > 7 are considered normal; 4 to 6, fairly low; and < 3 are generally regarded as critically low.
  scores on a scale | 8.95 (0.39) | 8.83 (0.38) | 8.89 (0.39)
Positive family history of allergic disease [Count of Participants; unit: Participants]
  No | 21 | 22 | 43
  Yes | 19 | 18 | 37
Positive family history of functional gastrointestinal diseases [Count of Participants; unit: Participants]
  No | 37 | 33 | 70
  Yes | 3 | 7 | 10
Clinical/surgical history [Count of Participants; unit: Participants]
  No prior clinical/surgical events were reported | 40 | 40 | 80
  Prior clinical/surgical events were reported | 0 | 0 | 0
Exposure to second-hand tobacco smoke within the home environment [Count of Participants; unit: Participants]
  No | 29 | 29 | 58
  Yes | 11 | 11 | 22
Smoking habits [Count of Participants; unit: Participants]
  Mother | 6 | 4 | 10
  Mother, Father | 3 | 1 | 4
  Father | 5 | 6 | 11
  No one | 26 | 29 | 55

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With >=50% Reduction in Mean Weekly Crying Duration
Description: Treatment success rate was evaluated in terms of reduction of crying duration, comparing mean weekly duration of the last Week (from T4 to T5) and mean weekly duration of Week 1 (from T0 to T1). The daily number and duration of crying episodes has been collected in the 'Evaluation of crying' section of the patient diary.
  Weekly mean is defined as the mean of the calculated average daily durations during the selected week and is described by means of descriptive statistics for continuous data. Mean changes from baseline (i.e. mean of the first Week) to the mean of the selected week will be computed as well.
  The following categories of patients has been defined:
  Success = patients who meet the criteria for the treatment success rate No Success = patients who do not meet the criteria for the treatment success rate Missing = patients who did not do the last visit (Visit T5 - at 28 days from baseline)
Time Frame: at 28 days from the baseline (Visit T5)
Population: Intention to Treat Set (ITT): all randomized patients who received at least one dose of study treatment. Following the intent-to-treat (ITT) principle, patients were analyzed according to the treatment they were assigned to at the randomization visit.
  Patients drop-out were also considered and classified as Treatment success rate = "Missing".
Measure: Count of Participants; unit: Participants
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
Participants
  Visit T5 - Success | 32 | 13
  Visit T5 - No Success | 3 | 24
  Visit T5 - Missing | 5 | 3
Statistical Analysis 1: Comparison: Bifidobacterium BB-12® vs Placebo; According to the results of a previous trial that looked at a probiotic's effect on infants with CI, it was estimated that when the sample size in each group is 33, the study has 80% power to detect an absolute difference of 35% in the treatment success rate (15% in the Placebo group and 50% in the treatment group) with a 0,05 alpha level. The number of infants that was included in the study was 80, with an expected maximum dropout rate of 20%; Test type: Other; p = 0.0001, Chi-squared

2. Secondary Outcome: Number of Crying Episodes
Description: Weekly mean of cries will be defined as the mean number of cries reported in the "Evaluation of behavior" section during the week (i.e. number of episodes/number of days with episodes) and will be described by means of descriptive statistics for continuous data.
  Mean changes from baseline (i.e. mean of the first Week) to the mean of the selected week will be analyzed too.
Time Frame: at 7 days (Visit T1 - baseline) and 28 days from the baseline (Visit T5)
Population: Intention to Treat Set (ITT): all randomized patients who received at least one dose of study treatment.
  The number of participants analyzed in Visit T5 is less then Visit T1 since 8 participants dropped from the study before Visit T5
Measure: Mean (Standard Deviation); unit: number of episodes
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
number of episodes
  Visit T1 - Baseline | 7.92 (2.79) | 8.28 (3.12)
  Visit T5: number analyzed (Participants) | 35 | 37
  Visit T5 | 3.15 (1.48) | 6.04 (2.42)
Statistical Analysis 1: Comparison: Bifidobacterium BB-12® vs Placebo; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Infectious Diseases Incidence
Description: Number of infections in respiratory system, gastrointestinal system, urinary tract and skin.
  An infection was defined as an Adverse Event with SOC equal to "Infections and Infestations".
Time Frame: at each visit, for 5 weeks starting from the enrollment in the study (Visit T0, T1, T2, T3, T4 and T5)
Population: Intention to Treat Set (ITT): all randomized patients who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: Number of infections
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
Number of infections | 0 (0) | 0 (0)

4. Secondary Outcome: Bowel Evacuation - Stool Frequency
Description: Daily frequency of bowel evacuation. The frequency of stools were collected daily in the diary. Stool frequency was evaluated as the mean of total daily stools reported per week.
Time Frame: at each weekly visit from baseline (Visit T1, T2, T3, T4 and T5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: daily number of bowel evacuations
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
daily number of bowel evacuations
  Visti T1 - Baseline | 5.30 (1.49) | 5.61 (1.60)
  Visit T2: number analyzed (Participants) | 40 | 39
  Visit T2 | 5.15 (1.63) | 5.50 (1.54)
  Visit T3: number analyzed (Participants) | 38 | 37
  Visit T3 | 4.92 (1.53) | 5.35 (1.45)
  Visit T4: number analyzed (Participants) | 37 | 37
  Visit T4 | 4.51 (1.51) | 5.10 (1.24)
  Visit T5: number analyzed (Participants) | 35 | 37
  Visit T5 | 4.34 (1.45) | 4.64 (1.23)
Statistical Analysis 1: Comparison: Bifidobacterium BB-12® vs Placebo; Test type: Other; p = 0.001, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Bowel Evacuation - Stool Consistency
Description: Stool consistency was evaluated as the number and the proportion of patients who reported at least one stool sample of each type per week, according to Bristol scale as follows:
  Type A = separate hard lumps, like nuts (hard to pass) Type B = sausage-shaped, but lumpy Type C = Like a sausage but with cracks on its surface Type D = like a sausage or snake, smooth and soft Only a descriptive statistics Type E = soft blobs with clear-cut edges (passed easily) Type F = fluffy pieces with ragged edges, a mushy stool Type G = watery, no solid pieces (entirely liquid). Patients could report more than one stool consistency per day then the sum of the "Count of Participants" for each group at each visit could be Greater then the "Overall Number of Participants Analyzed"
Time Frame: at each weekly visit from baseline (Visit T1, T2, T3, T4 and T5)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
participants
  T1: Patients with at least 1 stool of type C | 0 | 1
  T1: Patients with at least one stool of type D | 14 | 10
  T1: Patients with at least one stool of type E | 21 | 15
  T1: Patients with at least one stool of type F | 27 | 34
  T1: Patients with at least one stool of type G | 12 | 21
  T2: Patients with at least one stool of type C | 0 | 1
  T2: Patients with at least one stool of type D | 14 | 8
  T2: Patients with at least one stool of type E | 25 | 19
  T2: Patients with at least one stool of type F | 30 | 34
  T2: Patients with at least one stool of type G | 12 | 20
  T3: Patients with at least one stool of type C | 0 | 0
  T3: Patients with at least one stool of type D | 16 | 8
  T3: Patients with at least one stool of type E | 24 | 26
  T3: Patients with at least one stool of type F | 27 | 30
  T3: Patients with at least one stool of type G | 8 | 8
  T4: Patients with at least one stool of type C | 0 | 0
  T4: Patients with at least one stool of type D | 18 | 15
  T4: Patients with at least one stool of type E | 27 | 30
  T4: Patients with at least one stool of type F | 23 | 27
  T4: Patients with at least one stool of type G | 8 | 5
  T5: Patients with at least one stool of type C | 0 | 0
  T5: Patients with at least one stool of type D | 17 | 25
  T5: Patients with at least one stool of type E | 26 | 29
  T5: Patients with at least one stool of type F | 19 | 16
  T5: Patients with at least one stool of type G | 6 | 3

6. Secondary Outcome: Infant's Mood
Description: The infant's mood (calm, asleep, agitated, irritable) was collected daily in the diary and was evaluated as the number and the proportion of infants who reported at least one mood of each type per week.
  Patients could report more than one mood per day then the sum of the "Count of Participants" for each group at each visit could be greater then the "Overall Number of Participants Analyzed".
Time Frame: at each weekly visit from baseline (Visit T1, T2, T3, T4 and T5)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
participants
  T1: Pts with at least one mood equal to Calm | 4 | 5
  T1: Pts. with at least one mood equal to Asleep | 5 | 6
  T1: Pts. with at least one mood equal to Agitated | 38 | 25
  T1: Pts. with at least one mood equal to Irritable | 36 | 36
  T2: Pts. with at least one mood equal to Calm: number analyzed (Participants) | 40 | 39
  T2: Pts. with at least one mood equal to Calm | 14 | 7
  T2: Pts. with at least one mood equal to Asleep | 11 | 8
  T2: Pts. with at least one mood equal to Agitated | 37 | 32
  T2: Pts. with at least one mood equal to Irritable | 33 | 34
  T3: Pts. with at least one mood equal to Calm: number analyzed (Participants) | 38 | 37
  T3: Pts. with at least one mood equal to Calm | 28 | 12
  T3: Pts. with at least one mood equal to Asleep | 12 | 8
  T3: Pts. with at least one mood equal to Agitated | 34 | 33
  T3: Pts. with at least one mood equal to Irritable | 25 | 30
  T4: Pts. with at least one mood equal to Calm: number analyzed (Participants) | 37 | 36
  T4: Pts. with at least one mood equal to Calm | 35 | 15
  T4: Pts. with at least one mood equal to Asleep | 21 | 17
  T4: Pts. with at least one mood equal to Agitated | 32 | 36
  T4: Pts. with at least one mood equal to Irritable | 11 | 28
  T5: Pts. with at least one mood equal to Calm: number analyzed (Participants) | 35 | 37
  T5: Pts. with at least one mood equal to Calm | 35 | 17
  T5: Pts. with at least one mood equal to Asleep | 27 | 23
  T5: Pts. with at least one mood equal to Agitated | 9 | 34
  T5: Pts. with at least one mood equal to Irritable | 5 | 20

7. Secondary Outcome: Infant's Sleep
Description: Duration of sleep (in minutes) was collected daily in the diary during the entire study period. Mean daily duration of sleep by week was defined as the mean of the daily durations during the selected week and was described by means of descriptive statistics for continuous data.
Time Frame: at each weekly visit from baseline (Visit T1, T2, T3, T4 and T5)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
minutes
  Visit T1 - baseline | 678.14 (96.13) | 693.62 (121.79)
  Visit T2: number analyzed (Participants) | 40 | 39
  Visit T2 | 687.47 (113.41) | 696.68 (121)
  Visit T3: number analyzed (Participants) | 38 | 37
  Visit T3 | 722.37 (116.30) | 711.99 (128.87)
  Visit T4: number analyzed (Participants) | 37 | 36
  Visit T4 | 725.76 (112.54) | 725.14 (131.74)
  Visit T5: number analyzed (Participants) | 35 | 37
  Visit T5 | 713.20 (98.97) | 738.61 (141.58)

8. Secondary Outcome: Infant's Temper
Description: Duration of temper episodes (in minutes) was collected daily in the diary during the entire study period. Mean daily duration of temper episodes by week was defined as the mean of the daily durations during the selected week and was described by means of descriptive statistics for continuous data.
Time Frame: at each weekly visit from baseline (Visit T1, T2, T3, T4 and T5)
Population: Intention to Treat Set (ITT): all randomized patients who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
minutes
  Visit T1 - Baseline: number analyzed (Participants) | 20 | 19
  Visit T1 - Baseline | 158.82 (36.31) | 138 (34.71)
  Visit T2: number analyzed (Participants) | 21 | 18
  Visit T2 | 118.61 (45.59) | 117.24 (58.32)
  Visit T3: number analyzed (Participants) | 19 | 16
  Visit T3 | 89.48 (47.96) | 84.33 (46.76)
  Visit T4: number analyzed (Participants) | 17 | 16
  Visit T4 | 71.71 (54.79) | 84.89 (58.04)
  Visit T5: number analyzed (Participants) | 17 | 16
  Visit T5 | 36.79 (42.45) | 72.96 (40.22)

9. Secondary Outcome: Infant's Feeding
Description: Duration of feeding (in minutes) was collected daily in the diary during the entire study period. Mean daily feeding time by week was defined as the mean of the daily durations during the selected week and was described by means of descriptive statistics for continuous data.
Time Frame: at each weekly visit from baseline (Visit T1, T2, T3, T4 and T5)
Population: Intention to Treat Set (ITT): all randomized patients who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 40 | 40
minutes
  Visit T1 - Baseline: number analyzed (Participants) | 21 | 21
  Visit T1 - Baseline | 187.72 (35.95) | 177.72 (34.66)
  Visit T2: number analyzed (Participants) | 21 | 20
  Visit T2 | 186.13 (63.37) | 188.98 (32.75)
  Visit T3: number analyzed (Participants) | 20 | 19
  Visit T3 | 179.80 (55.16) | 185.98 (30.98)
  Visit T4: number analyzed (Participants) | 19 | 19
  Visit T4 | 180.31 (47.85) | 182.22 (28.70)
  Visit T5: number analyzed (Participants) | 18 | 19
  Visit T5 | 176.47 (38.55) | 182.26 (27.20)

10. Secondary Outcome: Calprotectin
Description: Evaluation of calprotectin levels in fecal samples
Time Frame: at 7 days (Visit T1 - baseline) and 28 days from the baseline (Visit T5)
Population: The analysis Population includes all participants for wich an evaluable fecal sample was available at Visit T1 and Visit T5
Measure: Mean (Standard Deviation); unit: mM/Kg
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 32 | 30
mM/Kg
  Visit T1 - Baseline | 667.76 (162.06) | 658.47 (112.61)
  Visit T5 | 802.64 (131.33) | 915.41 (106.47)

11. Secondary Outcome: Beta-defensin Type 2
Description: Evaluation of Beta-defensin type 2 levels in fecal samples
Time Frame: at 7 days (Visit T1 - baseline) and 28 days from the baseline (Visit T5)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 32 | 30
ng/g
  Visit T1 - baseline | 73.50 (10.92) | 69.41 (7.03)
  Visit T5 | 166.34 (43.79) | 127.97 (35.41)

12. Secondary Outcome: LL37 Peptide
Description: Evaluation of LL37 peptide levels in fecal samples
Time Frame: at 7 days (Visit T1 - baseline) and 28 days from the baseline (Visit T5)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/g
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 32 | 30
ng/g
  Visit T1 - Baseline | 5.50 (0.82) | 5.37 (0.83)
  Visit T5 | 7.65 (1.15) | 6.07 (1.41)

13. Secondary Outcome: Short Chain Fatty Acids - Butyrate
Description: Evaluation of Butyrate levels in fecal samples
Time Frame: at 7 days (Visit T1 - baseline) and 28 days from the baseline (Visit T5)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mM/Kg
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 32 | 30
mM/Kg
  Visit T1 - Baseline | 0.19 (0.14) | 0.17 (0.16)
  Visit T5 | 0.63 (0.49) | 0.32 (0.33)

14. Secondary Outcome: Secretory Immunoglobulin A (SIgA)
Description: Secretory immunoglobulin A (SIgA) levels in fecal samples
Time Frame: at 7 days (Visit T1 - baseline) and 28 days from the baseline (Visit T5)
Population: The analysis Population includes all the participants for wich an evaluable fecal sample was available at Visit T1 and Visit T5
Measure: Mean (Standard Deviation); unit: microg/g
Arm/Group | Bifidobacterium BB-12® | Placebo
Number analyzed (Participants) | 32 | 30
microg/g
  Visit T1 - Baseline | 84.79 (21.71) | 86.55 (12.13)
  Visit T5 | 250.65 (37.95) | 192.01 (27.12)

ADVERSE EVENTS:
Time Frame: 5 weeks starting from the patient enrollment
Arm/Group | Bifidobacterium BB-12® | Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bifidobacterium BB-12® (N=40) | Placebo (N=40)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03434249/SAP_000.pdf
  • Study Protocol (2019-12-04): https://cdn.clinicaltrials.gov/large-docs/49/NCT03434249/Prot_001.pdf